CLINICAL TRIAL: NCT01117454
Title: A Prospective Randomized Crossover Trial of Oral Flecainide for Catecholaminergic Polymorphic Ventricular Tachycardia
Brief Title: Flecainide for Catecholaminergic Polymorphic Ventricular Tachycardia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Prince Joseph Kannankeril, Principal Investigator, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 100472
Record Dates: First submitted 2010-05-04; First posted 2010-05-05 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Catecholaminergic Polymorphic Ventricular Tachycardia
Keywords: Catecholaminergic Polymorphic Ventricular Tachycardia; implantable cardioverter-defibrillator; flecainide
MeSH Terms: conditions — Polymorphic Catecholaminergic Ventricular Tachycardia | interventions — Flecainide; Adrenergic beta-Antagonists

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Flecainide then placebo (Other): In this crossover study, half of the subjects will be randomized to flecainide plus standard therapy with beta-blockers first, then crossover to placebo plus standard therapy with beta-blockers.
  Interventions: Drug: Flecainide Acetate; Drug: Placebo; Drug: Beta blocker
- Placebo then flecainide (Other): In this crossover study, half of the subjects will be randomized to placebo plus standard therapy with beta-blockers first, then crossover to flecainide plus standard therapy with beta-blockers.
  Interventions: Drug: Flecainide Acetate; Drug: Placebo; Drug: Beta blocker

INTERVENTIONS:
Drug: Flecainide Acetate — oral flecainide with the dose titrated to achieve a serum level between 0.5-0.8 mcg/ml
Drug: Placebo — placebo, similar in appearance to flecainide
Drug: Beta blocker — Standard therapy with beta-blocker (nadolol, atenolol, metoprolol, or propranolol) continues throughout the trial.

SUMMARY:
The purpose of this study is to test whether the addition of oral flecainide to standard therapy will reduce ventricular ectopy on exercise test compared to placebo plus standard therapy in patients with Catecholaminergic Polymorphic Ventricular Tachycardia.

DETAILED DESCRIPTION:
Catecholaminergic Polymorphic Ventricular Tachycardia (CPVT) is a genetic arrhythmia syndrome characterized by frequent ventricular ectopy and polymorphic, classically bidirectional ventricular tachycardia with physical or emotional stress, which also carries a risk of ventricular fibrillation and sudden death, despite no structural heart abnormality. Treatment consists of beta-blockers and/or calcium channel blockers, but up to 30% of patients require implantable cardioverter-defibrillators (ICDs) due to recurrent symptoms on medical therapy. In an animal model, flecainide was found to directly target the molecular defect in CPVT. In a retrospective clinical study in patients with CPVT we have seen improvement of ventricular ectopy on exercise tests when flecainide is added to standard therapy. We propose a prospective trial of flecainide added to standard therapy in CPVT patients to test the hypothesis that flecainide will reduce ventricular ectopy on exercise testing compared to placebo plus standard therapy.

This will be a single-blind (blinded subjects) randomized cross-over study, in which each patient will receive treatment A (flecainide or placebo) for at least 3 months and, after a 1 week wash-out, treatment B (placebo or flecainide) for at least 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of CPVT, based on:

   A. reproducible polymorphic or bidirectional ventricular tachycardia with exercise OR B. Ventricular ectopy on exercise test with RYR2 or CASQ2 mutation
2. Functioning ICD in place
3. On stable dose of standard therapy defined as the maximal tolerated dose of beta-blocker and may include a calcium channel blocker

Patients on flecainide or mexiletine are also eligible for enrollment after a 1 week "washout" period during which flecainide or mexiletine is discontinued, and standard therapy alone is used.

Exclusion Criteria:

1. Females who are pregnant or plan to be pregnant during the study period
2. Children < 5 years of age
3. Patients unable to perform treadmill exercise
4. Patients with significant structural heart disease
5. Patients with features consistent with Andersen-Tawil syndrome A. Periodic paralysis or unexplained weakness B. Dysmorphic facies C. Known KCNJ2 mutation
6. Patients with known hypersensitivity to flecainide
7. Patients on amiodarone
8. Patients not expected to comply with follow-up

Ages: 5 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prince J Kannankeril, MD, MSCI, Principal Investigator — Vanderbilt University
Locations (10):
- United States (10):
  - University of California Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - NYU Langone Medical Center, New York, New York
  - Duke University, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Vanderbilt University, Nashville, Tennessee
  - Cook Children's Hospital, Fort Worth, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Watanabe H, Chopra N, Laver D, Hwang HS, Davies SS, Roach DE, Duff HJ, Roden DM, Wilde AA, Knollmann BC. Flecainide prevents catecholaminergic polymorphic ventricular tachycardia in mice and humans. Nat Med. 2009 Apr;15(4):380-3. doi: 10.1038/nm.1942. Epub 2009 Mar 29. PMID 19330009
- [Background] van der Werf C, Kannankeril PJ, Sacher F, Krahn AD, Viskin S, Leenhardt A, Shimizu W, Sumitomo N, Fish FA, Bhuiyan ZA, Willems AR, van der Veen MJ, Watanabe H, Laborderie J, Haissaguerre M, Knollmann BC, Wilde AA. Flecainide therapy reduces exercise-induced ventricular arrhythmias in patients with catecholaminergic polymorphic ventricular tachycardia. J Am Coll Cardiol. 2011 May 31;57(22):2244-54. doi: 10.1016/j.jacc.2011.01.026. PMID 21616285
- [Background] Kannankeril PJ, Moore JP, Cerrone M, Priori SG, Kertesz NJ, Ro PS, Batra AS, Kaufman ES, Fairbrother DL, Saarel EV, Etheridge SP, Kanter RJ, Carboni MP, Dzurik MV, Fountain D, Chen H, Ely EW, Roden DM, Knollmann BC. Efficacy of Flecainide in the Treatment of Catecholaminergic Polymorphic Ventricular Tachycardia: A Randomized Clinical Trial. JAMA Cardiol. 2017 Jul 1;2(7):759-766. doi: 10.1001/jamacardio.2017.1320. PMID 28492868
- See also: Full text of publication in JAMA Cardiology — http://jamanetwork.com/journals/jamacardiology/fullarticle/2626499

RESULTS

PARTICIPANT FLOW:
Groups:
- Flecainide Then Placebo: In this crossover study, half of the subjects will be randomized to flecainide plus standard therapy first, then crossover to placebo plus standard therapy.
  flecainide: oral flecainide will be added to standard therapy with the dose titrated to achieve a serum level between 0.5-0.8 mcg/ml
- Placebo Then Flecainide: In this crossover study, half of the subjects will be randomized to placebo plus standard therapy first, then crossover to flecainide plus standard therapy.
  flecainide: oral flecainide will be added to standard therapy with the dose titrated to achieve a serum level between 0.5-0.8 mcg/ml
Period: Overall Study
Arm/Group | Flecainide Then Placebo | Placebo Then Flecainide
Started | 6 | 8
Completed | 6 | 7
Not Completed | 0 | 1
Not completed — Pregnancy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Flecainide Then Placebo | Placebo Then Flecainide | Total
Number analyzed (Participants) | 6 | 8 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 7 | 10
  Between 18 and 65 years | 3 | 1 | 4
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Ventricular Ectopy or VT During Exercise Treadmill Testing
Description: Hypothesis: the addition of oral flecainide to standard therapy will reduce ventricular ectopy and/or VT on treadmill exercise treadmill testing in patients with CPVT, compared to placebo plus standard therapy.
Time Frame: 3 months
Population: 1 participant did not complete treadmill test
Measure: Count of Participants; unit: Participants
Groups:
- Flecainide: All participants when receiving flecainide
- Placebo: All participants when receving placebo
Arm/Group | Flecainide | Placebo
Number analyzed (Participants) | 12 | 12
Participants | 2 | 9
Statistical Analysis 1: Comparison: Flecainide vs Placebo; Test type: Superiority; p = 0.008, Wilcoxon (Mann-Whitney); Wilcoxon signed rank with continuity correction

ADVERSE EVENTS:
Time Frame: Participants were followed for the duration of the study, an average of 26 months
Arm/Group | Flecainide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 2/13 | 2/13
Other Adverse Events (participants affected / at risk) | 11/13 | 6/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flecainide (N=13) | Placebo (N=13)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Implantable Cardioverter-Defibrillator Infection (Cardiac disorders) | 0 (0) | 1 (1)
Back pain requiring Surgery (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Allergic Reaction requiring Hospitalization (Immune system disorders) | 1 (1) | 0 (0)
Supraventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Vasovagal Syncope (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flecainide (N=13) | Placebo (N=13)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Musculoskelatal Injury (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
lightheadedness (Nervous system disorders) | 1 (1) | 0 (0)
palpitations (Cardiac disorders) | 0 (0) | 2 (2)
dizziness (Nervous system disorders) | 2 (2) | 0 (0)
phantom shock (Psychiatric disorders) | 0 (0) | 1 (1)
anorexia (Gastrointestinal disorders) | 1 (1) | 0 (0)
fatigue (General disorders) | 1 (1) | 0 (0)
blurry vision (Eye disorders) | 4 (5) | 0 (0)
constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
influenza (Infections and infestations) | 1 (1) | 0 (0)
insominia (General disorders) | 1 (1) | 0 (0)
left side pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes